CLINICAL TRIAL: NCT04200807
Title: Non-invasive Measurement of Neonatal Central and Peripheral Hemodynamics, as Valuable Diagnostic and Treatment Efficiency Criterium of Neonatal Sepsis
Brief Title: Non-invasive Measurement of Neonatal Central and Peripheral Hemodynamics
Acronym: NInHeDyNeo
Status: Completed | Type: Observational
Sponsor: Vilnius University (Other)
Responsible Party: Sponsor
Other Study IDs: NCPKV-2017
Record Dates: First submitted 2019-11-18; First posted 2019-12-16 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2020-09

CONDITIONS: Pre-Term; Neonatal Infection
Keywords: cardiac output; echocardiography; USCOM; neonates
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy preterm neonate: Neonate 26 weeks to 36 weeks + 6 days of gestation, without congenital heart defects and/or hemodynamically significant fetal circulation, any respiratory therapy, nor need of supplemental oxygen. Subjects had no clinically and laboratory-identified infections.
  Interventions: Device: Ultrasound Cardiac Output Monitor (USCOM 1A)
- Healthy term neonate: Neonate from 37 weeks of gestation, without congenital heart defects and/or hemodynamically significant fetal circulation, any respiratory therapy, nor need of supplemental oxygen. Subjects had no clinically and laboratory-identified infections.
  Interventions: Device: Ultrasound Cardiac Output Monitor (USCOM 1A)
- Sick neonate: Neonate of any gestation, without congenital heart defects, with clinically and laboratory-identified infection.
  Interventions: Device: Ultrasound Cardiac Output Monitor (USCOM 1A)

INTERVENTIONS:
Device: Ultrasound Cardiac Output Monitor (USCOM 1A) — doplerometry with USCOM and echocardiograph is made for assessing central blood flow and spectroscopy with NONIN- for the blood flow in individual peripheral organs (brain and kidney)
  Other Names: GE LOGIQ S8 XDclear 2.0 ultrasound system with S4-10-D (3-9MHz) probe; NONIN Equanox near-infrared spectroscope

SUMMARY:
Non-invasively neonatal cardiac output can be measured by multiple methods, but the gold standard still remains conventional echocardiography. It is accurate, but needs a long training for new users to assess cardiac function. Continuous-wave Doppler ultrasound monitor USCOM is a relatively new monitor which can perform faster and less complex cardiac function measurement, also it is easier for the operator to get trained. The aim of the study is to assess the level of agreement between cardiac output measured with conventional echocardiography and with USCOM, to present normal ranges for neonates of different gestational age and to look for early signs of hemodynamic changes during sepsis.

ELIGIBILITY:
Inclusion Criteria:

* newborns of any gestational age
* parental consent acquired

Exclusion Criteria:

* congenital malformations
* hemodynamic instability in control group
* any respiratory support in control group
* infection in control group

Ages: 26 Weeks to 44 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study enrolled both preterm and full-term newborns of any gestational age, without congenital heart defects and/or hemodynamically significant fetal circulation, any respiratory therapy, nor need of supplemental oxygen. Subjects had no clinically and laboratory-identified infections in control group.
Sampling Method: Non-Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2017-09-12 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Weight measurement | 1 minute
  weight in grams
Height measurement | 1 minute
  length in centimeters
Chest and head circumference | 1 minute
  Chest and head circumference in centimeters
Blood pressure measurement | 1 minute
  non- invasive arterial blood pressure measurement in mmHg
Pulse rate measurement | 1 minute
  pulse rate in beats per minute
Near- Infrared Spectroscopy for regional blood flow | 15-20 minutes
  One sensor on the forehead, another- on the back to check for regional blood flow in the brain and kidney with Near- Infrared Spectroscopy
Echocardioscopy for left ventricular outflow tract diameter | 2-3 minutes
  Echocardiography for left ventricular outflow tract diameter in centimeters
Echocardioscopy to measure velocity time integral | 3 minutes
  Echocardiography to measure velocity time integral at the aortic valve in centimeters. After that the software of the device calculates cardiac output.
USCOM examination | 3-5 minutes
  USCOM 1A uses continuous wave Doppler for flow curves, which are obtained at the suprasternal notch for an optimal flow signal at the aortic valve. The software of the device calculates cardiac output then

CONTACTS AND LOCATIONS:
Overall Officials: Vytautas Usonis, MD, Study Director — Vilnius University
Locations (1):
- Vilnius University, Neonatology Centre, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pliauckiene A, Liubsys A, Vankeviciene R, Usonis V. Ultrasonic cardiac output monitor provides effective non-invasive bedside measurements of neonatal cardiac output. J Clin Monit Comput. 2022 Jun;36(3):803-807. doi: 10.1007/s10877-021-00711-2. Epub 2021 Apr 30. PMID 33929641